CLINICAL TRIAL: NCT01903044
Title: Multicentric Study of the Autologous Bone Marrow-derived Mononuclear Cells Injection for Treatment of the Patients With Critical Lower Extremity Ischemia
Brief Title: Safety and Efficacy of Autologous Bone Marrow Stem Cells for Lower Extremity Ischemia Treating
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pontifícia Universidade Católica do Paraná (Other)
Collaborators: Instituto de Moléstias Cardiovasculares de São José do Rio Preto, Brazil (Unknown); Hospital Sao Rafael (Other); Hospital Geral Nacional Enrique Cabrera, Cuba (Unknown); Instituto de Hematología e Inmunología, Cuba (Unknown); Fundação Araucária (Other)
Responsible Party: Principal Investigator, Alexandra Cristina Senegaglia, PhD, Pontifícia Universidade Católica do Paraná
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMI_ 404732/2012-7
Record Dates: First submitted 2013-07-10; First posted 2013-07-19 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Lower Extremity Ischemia; Leg Ulcer; Peripheral Vascular Disease; Diabetic Foot; Gangrene
Keywords: Lowe extremity ischemia; Bone marrow; Neoangiogenesis
MeSH Terms: conditions — Leg Ulcer; Peripheral Vascular Diseases; Diabetic Foot; Gangrene; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BM-MNC injection (Experimental): Injection of autologous bone marrow-derived mononuclear cells
  Interventions: Procedure: BM-MNC injection

INTERVENTIONS:
Procedure: BM-MNC injection — BM-MNC cells will be injected in aliquots of 1 ml at multiple regions of the leg muscles

SUMMARY:
The purpose of this study is to determine whether autologous bone marrow-derived stem cells are effective in the treatment of lower extremity ischemia.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) is a debilitating and disabling disease. Symptoms include pain at rest, loss of tissue integrity, distal amputations and have a major impact on the quality of life. Despite recent advances in surgical vascular procedures, a large number of patients (approximately 40%) are not eligible for these revascularization procedures. New strategies for revascularization need to be explored. Besides, in some cases results of such interventions do not give desirable effect, search of new methods of treatment therefore is necessary. Recent evidence indicates that bone marrow-derived mononuclear cells (BM-MNC) are a potential new therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

* Critical lower limb ischemia, defined as ischemic pain at rest and / or the presence of minor tissue loss, with the possibility of healing.
* Failure of conventional medical treatment and attempts to open or percutaneous revascularization before, with an observation period of two months after the last attempt at revascularization.
* Patients considered at high risk for new revascularization procedure by at least two independent observers.

Exclusion Criteria:

* Expected life span less than six months
* Large tissue loss in the ischemic limb indicating the need for limb amputation in the short term.
* Evidence of osteomyelitis in the ischemic extremity.
* Current or previous history of neoplasia.
* Unstable angina, recent stroke or other medical condition that contraindicate anesthesia for bone marrow aspiration.
* Proliferative retinopathy.
* Debilitating disease with a life span less than one year.
* Myelofibrosis, myelodysplasia or other diseases that affect the bone marrow.
* Use of alcohol in excess of twice-daily doses or history of illicit drug use.
* Need for continuous high doses of drug therapy with steroids (more than 7.5 mg/day).
* Positivity for HIV or syphilis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Wound healing (wound size, wound stage) - monitoring the healing of trophic lesions | 3 months

SECONDARY OUTCOMES:
Clinical outcome classification | 3 months, 6 months
  Improvement of symptoms, functional capacity, exercises tolerance assessed by change in Rutherford scale of CLI
Pain and analgesics use | 3 months
Quality of life outcome | 3 months, 6 months
Improvement of the coronary and collateral circulation. | 3 months
Survival without amputation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Brofman, PhD, Principal Investigator — Pontifícia Universidade Católica do Paraná
Locations (1):
- Pontifícia Universidade Católica do Paraná, Curitiba, Paraná, Brazil